CLINICAL TRIAL: NCT04328883
Title: A Phase 1, Single-dose, Open-label, Pilot Study to Compare the Pharmacodynamics and Pharmacokinetics of Acetylsalicylic Acid Inhalation Powder With Non-Enteric-Coated Chewable Aspirin in Healthy Adults
Brief Title: Pharmacodynamics and Pharmacokinetics of Aspirin Inhalation Powder With Non-Enteric-Coated Chewable Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InovaHCS
Record Dates: First submitted 2019-12-09; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-12

CONDITIONS: Platelet Aggregation Inhibitors
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 162 mg Non-Enteric-Coated Chewable aspirin (Active Comparator): Non-enteric coated aspirin (162mg, single dose)
  Interventions: Drug: Aspirin
- 50 mg ASA inhalation powder (Experimental): Dry powder inhaled aspirin (50mg,1 dry powder inhalation capsule using dry powder inhaler, single dose)
  Interventions: Drug: Aspirin
- 100 mg ASA inhalation powder (Experimental): Dry powder inhaled aspirin (100mg,1 dry powder inhalation capsule using dry powder inhaler, single dose)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Oral and inhaled ASA formulations
  Other Names: Bayer Aspirin

SUMMARY:
ASA inhalation powder is an inhaled nonsteroidal anti-inflammatory drug-device combination that has been developed to reduce the risk of vascular mortality in patients with suspected acute myocardial infarction (MI), an FDA approved indication for oral formulations of aspirin.

The primary goal of study OTP-P0-926 is to collect pharmacokinetic (PK)and pharmacodynamics (PD) pilot data to determine onset and extent of aspirin response after administration of varying doses of inhaled ASA (50-100mg) and 162 mg Non-Enteric-Coated Chewable ASA. PD will be assessed using standard methods to measure platelet inhibition by aspirin including platelet aggregation, serum thromboxane,and urinary thromboxane. Furthermore, the pharmacokinetics (PK) of ASA will be determined and compared to PD measurements. Results of this pilot study will guide dosing in a subsequent larger Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-55 years of age
* Non-smokers
* Body mass index (BMI) within 18.5 kg/m2 to 32.0 kg/m2
* Female subjects of childbearing potential must agree to use acceptable methods of birth control or abstain from sex during study participation and must have a negative serum or urine pregnancy test
* Subjects must be healthy as determined by medical history, physical examination, vital signs, and clinical laboratory evaluation
* Signed informed consent

Exclusion Criteria:

* At screening visit, subjects with a forced expiratory volume in 1 second (FEV1) (i.e., FEV1% predicted < 80%).
* At screening visit, subjects with a forced expiratory flow at 25%-75% (FEF 25%-75%) of pulmonary volume < 70% predicted.
* Patients with a flow rate <70 L/min with a G-16 training device set at medium resistance.
* Hematocrit value ≤32%
* Clinically significant hemoglobin value, at screening, as per investigator.
* Arachidonic acid induced-maximum platelet aggregation <50%.
* Platelet count <142,000 or > 450,000 µL.
* Presence of any tongue piercings or history of any tongue piercings in the last 90 days prior to the first study drug administration.
* Presence of braces, partials or dentures.
* Clinically significant abnormal laboratory parameters.
* Antiplatelet agents (ASA, NSAID's, P2Y12 inhibitors, etc.) within 10 days of dosing visit.
* HIV, hepatitis B or C infection.
* Presence of clinically significant cardiovascular, pulmonary, hepatic, renal, endocrinological, hematological, immunologic, metabolic, neurological, or gastrointestinal disease.
* Clinically significant physical examination.
* History of hypersensitivity or allergy to aspirin.
* History of significant bleeding disorders.
* History of peptic ulcer disease.
* History of asthma or chronic obstructive pulmonary disease.
* Concurrent corticosteroid use with the exception of topical; any previous use must have occurred at least 90 days prior to Day 1 of the study and be approved by the Investigator.
* Administration of any prescription/over the counter medications/herbal/nutritional supplements within 14 days that has an effect on platelets prior to visit1 of the study.
* Administration of any investigational drug product (IP) within 30 days prior to visit 1.
* ALT ≥ 3xULN.
* Total Bilirubin > 1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Donation of blood or platelets within 60 days prior to visit 1.
* Any condition, illness, or disease that in the opinion of the investigator would interfere with the subject's ability to comply with the requirements of this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Compare the onset and extent of the pharmacodynamic effect of ASA inhalation powder (50-100 mg) and chewed non-enteric coated aspirin (162 mg) on arachidonic acid (AA)-induced platelet aggregation. | 24 hours
  Change from pre-dose in 1mM arachidonic-induced platelet aggregations at 2, 5, 10, 20,30, 40 minutes and 1,4, and 24hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.

SECONDARY OUTCOMES:
Compare the onset and extent of the pharmacodynamic effect of ASA inhalation powder and chewed non-enteric coated aspirin on ADP-induced platelet aggregation. | 24 hours
  Change from pre-dose on 5uM ADP-induced platelet aggregation at 2, 5, 10, 20,30, 40 minutes and 1,4, and 24hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.
Compare the onset and extent of the pharmacodynamic effect of ASA inhalation powder and chewed non-enteric coated aspirin on Collagen-induced platelet aggregation. | 24 hours
  Change from pre-dose on 4ug Collagen-induced platelet aggregation at 2, 5, 10, 20,30, 40 minutes and 1,4, and 24hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.
Compare the onset and extent of the pharmacodynamic effect of ASA inhalation powder and chewed non-enteric coated aspirin on serum concentrations of thromboxane B2 (TxB2). | 24 hours
  Change from pre-dose on serum concentrations of TxB2 at 2, 5, 10, 20,30, 40 minutes and 1,4, and 24hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.
Compare the onset and extent of the pharmacodynamic effect of ASA inhalation powder and chewed non-enteric coated aspirin on 6-keto- PGI1α. | 24 hours
  Change from pre-dose on 6-keto- PGI1α at 2, 5, 10, 20,30, 40 minutes and 1,4, and 24hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.
Compare the extent of the pharmacodynamic effect of ASA inhalation powder and chewed non-enteric coated aspirin on urinary 11-dehydro TxB2. | 24 hours
  Change from pre-dose on urinary 11-dehydro TxB2 at 4, and 24 hours after dosing with 50, 100mg aspirin dry powder inhalation and 162mg chewed non-enteric coated aspirin.
Compare the time to maximum drug concentration (Tmax) on ASA and salicylic acid (SA) pharmacokinetics following single doses of ASA inhalation powder and oral (Non-Enteric-Coated Chewable ) aspirin | 24 hours
  Compare Tmax between treatment groups
Compare the maximum drug concentration (Cmax) on ASA and salicylic acid (SA) pharmacokinetics following single doses of ASA inhalation powder and oral (Non-Enteric-Coated Chewable ) aspirin | 24 hours
  Compare Cmax between treatment groups
Evaluate change in forced expiratory-1 (FEV-1) after a single dose of acetylsalicylic acid (ASA) inhalation powder administered as ASA inhalation powder | 24 hours
  Evaluate change in forced expiratory-1 (FEV-1) from pre-dose measures after a single dose of acetylsalicylic acid (ASA) inhalation powder administered as ASA inhalation after 4 and 24hours post dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurbel PA, Bliden KP, Tantry US. Defining platelet response to acetylsalicylic acid: the relation between inhibition of serum thromboxane B2 and agonist-induced platelet aggregation. J Thromb Thrombolysis. 2021 Feb;51(2):260-264. doi: 10.1007/s11239-020-02334-x. Epub 2020 Nov 10. PMID 33170486